CLINICAL TRIAL: NCT00110383
Title: Effectiveness of School Based Supervised Asthma Therapy
Brief Title: Comparison of School-Based Supervised Versus Parental Supervised Asthma Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Lynn B. Gerald, PhD, MSPH, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 174; R01HL075043 (NIH)
Record Dates: First submitted 2005-05-06; First posted 2005-05-09 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2007-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Supervised therapy
  Interventions: Behavioral: School-Based Supervised Asthma Therapy
- 2 (No Intervention): Inhaled steroid use as usual care

INTERVENTIONS:
Behavioral: School-Based Supervised Asthma Therapy — Child's inhaled steroid use supervised daily at school
  Arms: 1

SUMMARY:
1. Develop a simple school-based intervention using school-based supervised asthma therapy to increase adherence to asthma medication.
2. Implement a school-based internet monitoring system within both the school-based supervised asthma therapy and parent supervised asthma therapy groups to record asthma symptoms, peak flow meter readings, school absences, and usage of rescue medications at school.
3. Randomly assign 250 children from inner-city school systems to either school-based supervised asthma therapy or parental supervised asthma therapy.
4. Compare children assigned to school-based supervised asthma therapy with children assigned to parent supervised asthma therapy, in regards to time-averaged proportion having at least one exacerbation per month, rescue medication use, peak flow meter readings, asthma symptoms, school absences, and asthma self-management knowledge.

DETAILED DESCRIPTION:
BACKGROUND:

Pediatric asthma is a well-documented public health issue in the United States. The impact of pediatric asthma can be measured by both health care costs and morbidity. Whereas many factors contribute to the high health care costs of asthma, much of the morbidity can be directly attributed to lack of adherence to medical treatments. The consequence of non-adherence for most individuals with ashtma is exacerbations. Greater numbers of exacerbations lead to increased school absenteeism, greater activity limitations, decreased quality of life for both parent and child, increased urgent health care use and costs, and increased parental days missed at work. Therefore, adherence to treatment is essential for proper asthma management and ultimate reductions in morbidity.

Asthma morbidity, as measured by the number of exacerbations, is largely preventable with patient education and optimal treatment. However, it has been demonstrated that patient education alone is insufficient to decrease asthma morbidity. Optimal treatment is essential to control asthma morbidity. Inhaled corticosteroids offer considerable protection against asthma exacerbations. However, only a minority of asthma patients take their inhaled steroids as recommended by the National Asthma Education and Prevention Program (NAEPP) guidelines. Therefore, the Pediatric Asthma Guidelines recommend development and testing of programs (including school-based programs) to increase adherence with therapy.

Because morbidity is higher in inner-city, low-income, minority children, this study will collaborate with several inner-city, low-income, minority school districts to examine the effects of school-based supervised asthma therapy.

DESIGN NARRATIVE:

This study is a longitudinal two-group trial of the effectiveness of a school-based supervised asthma therapy program. Two hundred and fifty children will be randomly assigned to one of two groups: school-based supervised asthma therapy or parental supervised asthma therapy. The children will be followed for 16 months.

ELIGIBILITY:
Inclusion Criteria:

* Persistent asthma requiring daily controller medication
* Enrolled at a participating elementary school

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 295 (Actual)
Dates: Start 2004-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbations | Measured at 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynn B. Gerald, PhD, MSPH, Study Chair — University of Alabama Birmingham Lung Health Center
Locations (1):
- University of Alabama Birmingham Lung Health Center, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Gerald LB, Gerald JK, Gibson L, Patel K, Zhang S, McClure LA. Changes in environmental tobacco smoke exposure and asthma morbidity among urban school children. Chest. 2009 Apr;135(4):911-916. doi: 10.1378/chest.08-1869. Epub 2008 Nov 18. PMID 19017893